CLINICAL TRIAL: NCT00372736
Title: A Phase I Study of AEG35156 Given as a 2 Hour Intravenous Infusion in Combination With Docetaxel in Patients With Solid Tumours
Brief Title: AEG35156 and Docetaxel in Treating Patients With Locally Advanced, Metastatic, or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I166B; CAN-NCIC-IND166B (Other: PDQ); CDR0000486837 (Other: PDQ)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — AEG 35156; Docetaxel; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: AEG35156 — After a recommended phase II dose (RPTD) of AEG35156 has been determined with docetaxel 75 mg/m2, patients will be accrued to the RPTD-1 plus docetaxel 100 mg/m2, and possibly RPTD plus docetaxel 100 mg/m2, to determine the RPTD of AEG35156 in combination with docetaxel 100 mg/m2 given every three weeks.
Drug: docetaxel — After a recommended phase II dose (RPTD) of AEG35156 has been determined with docetaxel 75 mg/m2, patients will be accrued to the RPTD-1 plus docetaxel 100 mg/m2, and possibly RPTD plus docetaxel 100 mg/m2, to determine the RPTD of AEG35156 in combination with docetaxel 100 mg/m2 given every three weeks.
Genetic: protein expression analysis — Cycle 1: Pre-dose on Days -2, 1, 8 and 15; repeat every 2-4 days if LFTs > 5 x ULN1 Cycle 2: Prior to each infusion; repeat every 2-4 days if LFTs > 5 x ULN1
Genetic: reverse transcriptase-polymerase chain reaction — Data will be summarized by descriptive statistics relevant to each of the proposed pharmacodynamic studies.
Other: flow cytometry — Data will be summarized by descriptive statistics relevant to each of the proposed pharmacodynamic studies.
Other: immunoenzyme technique — Data will be summarized by descriptive statistics relevant to each of the proposed pharmacodynamic studies.
Other: immunohistochemistry staining method — The plasma concentration/ time data will be analysed using non-compartmental methods. The pharmacokinetic parameters to be determined for AEG35156 include the maximum observed plasma concentration (Cmax), the half-life (T1/2), and mean residence time (MRT).
Other: laboratory biomarker analysis — The plasma concentration/ time data will be analysed using non-compartmental methods. The pharmacokinetic parameters to be determined for AEG35156 include the maximum observed plasma concentration (Cmax), the half-life (T1/2), and mean residence time (MRT).

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. AEG35156 may help docetaxel work better by making tumor cells more sensitive to the drug.

PURPOSE: This phase I trial is studying the side effects and best dose of AEG35156 when given together with docetaxel in treating patients with locally advanced, metastatic, or recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and define a recommended phase II dose of AEG35156 in combination with docetaxel in patients with locally advanced, metastatic, or recurrent solid tumors.

Secondary

* Determine the qualitative and quantitative toxicities of AEG35156 in combination with docetaxel given and define the duration and reversibility of those toxicities.
* Determine the pharmacokinetic profile of this regimen.
* Assess, preliminarily, the antitumor activity of this regimen in these patients.
* Assess the pharmacodynamic effects of AEG35156 on X-linked inhibitor of apoptosis levels and apoptosis in peripheral blood mononuclear cells and in tumor tissue of these patients.
* Evaluate M30/M65 cytokeratin 18 level (a marker of apoptosis/necrosis of epithelial tumors) in serum of these patients.

OUTLINE: This is a multicenter, open-label, dose-escalation study of AEG35156.

Patients receive AEG35156 IV over 2 hours on days -1, 0, 1, 8, and 15 during course 1 and on days 1, 8, and 15 of all subsequent courses. Patients also receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AEG35156 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which ≥ 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients receive AEG35156 at the recommended phase II dose (RPTD).

Blood is drawn periodically for pharmacokinetic and pharmacodynamic studies. Samples are examined by flow cytometry, immunoenzyme methods, and reverse transcriptase-polymerase chain reaction for biological markers. Tumor tissue (archival and fresh) is collected from patients treated at the RPTD and examined by immunohistochemical methods and biological marker analysis.

After completion of study treatment, all patients are followed at 4 weeks. Patients with response or stable disease ongoing are followed every 3 months thereafter until relapse/progression. Patients with protocol-related toxicity also followed q 3 months until resolution to ≤ grade 2.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Locally advanced, metastatic, or recurrent disease that is refractory to standard curative therapy or for which no curative therapy exists
* Clinically and/or radiologically documented disease
* Treatment with single-agent docetaxel is a reasonable treatment option
* No newly diagnosed CNS metastases

  * Previously treated and stable (≥ 6 months) intracranial disease allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* PT or INR and PTT normal
* Creatinine normal
* Bilirubin normal
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Gamma-glutamyl transferase ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No underlying serious illness or medical condition that might be aggravated by treatment or might interfere with study treatment, including, but not limited to, the following:

  * Serious uncontrolled infection
  * Significant cardiac dysfunction
  * Significant neurological disorder that would impair the ability to obtain informed consent
* No known bleeding disorders
* No prior serious allergic reaction to taxane (paclitaxel or docetaxel)
* No pre-existing peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy and recovered
* At least 2 weeks since prior hormonal therapy or immunotherapy
* At least 4 weeks since prior external-beam radiotherapy to < 30% of marrow-bearing areas

  * Low-dose, nonmyelosuppressive radiotherapy allowed
* At least 2 weeks since prior surgery and recovered
* More than 4 weeks since prior investigational agents or new anticancer therapy
* No prior nephrectomy
* No other concurrent chemotherapy
* No concurrent radiotherapy

  * Small-volume, non-myelosuppressive palliative radiotherapy allowed
* No other concurrent experimental drugs or anticancer therapy
* No concurrent therapeutic dose anticoagulant therapy

  * Non-therapeutic dose anticoagulant therapy (i.e., 1 mg daily oral warfarin) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-07-27 (Actual); Primary Completion 2009-03-24 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of AEG35156 in combination with docetaxel | 2-3 years
  Doses of AEG35156 escalated as shown in protocol section 4.3 in patient cohorts given a fixed dose of docetaxel. MTD defined as that dose level at which ≥ 2/6 patients experienced DLT (as defined in protocol section 4.6)
Recommended phase II dose | 2-3 years
  RPTD for AEG35156 defined as one dose lower than MTD

SECONDARY OUTCOMES:
Toxicities | Every 3 weeks
  Toxicities evaluated according to NCI CTCAE v3.0
Pharmacokinetic profile | Each cycle
  Venous blood samples for determination of AEG35156 concentration obtained on all patients during cycle 1 and 2 as per protocol section 17.2
Antitumor activity | Every 6 weeks
  All patients with measurable disease at baseline evaluated for response using RECIST criteria as described in protocol section 10.0
Pharmacodynamic effects of AEG35156 on X-linked inhibitor of apoptosis levels and apoptosis in peripheral blood mononuclear cells and tumor tissue | Each cycle
  Venous blood samples collected for PD studies as described in protocol Section 17.0. Fresh tissue biopsies also collected in patients entered at the RPTD.
M30/M65 cytokeratin 18 level | Each cycle
  Venous blood samples collected for determination of M30/M65 cytokeratin 18 and nucleosomal DNA as described in protocol section 17.0

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, MD, Study Chair — McGill Cancer Centre at McGill University
Locations (3):
- Canada (3):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No